CLINICAL TRIAL: NCT04036786
Title: Evaluation of the Education and Counseling Program on Pregnant Women With Risk of Preeclampsia: A Prospective Randomized Controlled Trial
Brief Title: Education and Counseling Program on Pregnant Women With Risk of Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Meltem Ugurlu, Assistant Proffessor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05555807841
Record Dates: First submitted 2019-07-18; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy
Keywords: pre-eclampsia; pregnancy; healthy lifestyle; self efficacy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study was a single-center, single-blinded, prospective randomized controlled trial (RCT), parallel-group RCT comparing the effects of a preeclampsia education and counseling program during pregnancy with standard antenatal care. Participants were 132 pregnant women with risk of preeclampsia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study gorup (Experimental): The study was a prospective randomized trial with a control group (standard care group) and an intervention group, using a repeated measures design. Sixty six pregnant participants with preeclampsia risk were included in the control group and 66 pregnant participants with preeclampsia risk were included in the intervention (exercise) group.
  Interventions: Behavioral: study group
- control group (Other): The study was a prospective randomized trial with a control group (standard care group) and an intervention group, using a repeated measures design. Sixty six pregnant participants with preeclampsia risk were included in the control group and 66 pregnant participants with preeclampsia risk were included in the intervention (exercise) group.
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: study group — We prepared a preeclampsia education booklet in accordance with the literature,The content of the booklet was guided by the opinion of experts. It was written in easily understandable language and contained attractive and colorful illustrations. This booklet contents were definition and risk factors for the development of preeclampsia, maternal and fetal damages, recommendations for preventing its development (diet, rest, study, exercise, coping with stress techniques), follow-up of symptoms at home (blood pressure, weight and edema follow-up, counting fetal movements), danger signs, drug use, follow up in hospital, risk of developing in subsequent pregnancies, and its results. Pregnant women in the study group were given education and counseling at four times in addition to standard care, using the preeclampsia education booklet, in a special place. The participants' questions were answered, and each received a copy of the booklet.
  Arms: study gorup
Behavioral: standard care — standard pregnancy follow up
  Arms: control group

SUMMARY:
The aim of the study is to evaluate the effect of education and counseling program on healthy lifestyle behaviors, self-efficacy and maternal/neonatal consequences of pregnant women with risk of preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia affects 3% to 5% of pregnancies, and is a pregnancy-specific syndrome; it leads to maternal, fetal and neonatal morbidity and mortality worldwide especially in developing countries. If not treated, pregnant woman may have many serious complications, such as pulmonary edema, eclampsia, stroke, placental abruption, and acute renal diseases . Babies born to mothers with preeclampsia have an increased risk of low Apgar scores, neonatal encephalopathy, seizures, neonatal intensive care admission, and neonatal deaths caused by preterm birth and low gestational age. Preeclampsia also affects the health-related quality of life negatively.

Since the etiology and pathogenesis of preeclampsia is unclear, it is very important to investigate the risk factors of preeclampsia to identify the pregnant women in the risk group, and to ensure more intensive care, observation and follow-ups. The known risk factors for preeclampsia include primiparity, advanced maternal age, family history of preeclampsia, previous preeclamptic pregnancy, autoimmune diseases, hypertension, history of thrombophilia, diabetes, in vitro fertilization, multifetal pregnancy, type I diabetes mellitus or type II diabetes mellitus and obesity..

It is known that the population has difficulty understanding even basic information related to health, and especially preeclampsia. Increasing the preeclampsia knowledge of women will help them to recognize early symptoms, and negative signs of preeclampsia, and may lead them to seek earlier individual care. Also, it is estimated that appropriate patient education and counseling for preeclampsia may prevent half of the most serious consequences related to maternal symptoms. This estimation is supported by a study, that women diagnosed with preeclampsia receiving proper and timely follow-up had fewer adverse events than those with delayed diagnosis. Preeclampsia education and counseling subjects may include recommendations for increasing awareness (preeclampsia signs and signs of danger, follow-up at home) and lifestyle modifications (physical activity, coping with stress, nutrition advices) to contribute to the prevention preeclampsia risks.

Although many studies have been carried out on medical treatment and improved outcomes in women with preeclampsia, there are limited studies about the consequences of education and counseling of pregnant women with risk of preeclampsia. Therefore, the objective of this study was to evaluate the effects of maternal and neonatal consequences of an education and counseling program on at-risk pregnant women.

Trial Design and Participants This study was a single-center, single-blinded, prospective randomized controlled trial (RCT), parallel-group RCT comparing the effects of a preeclampsia education and counseling program during pregnancy with standard antenatal care. Participants were 132 pregnant women with risk of preeclampsia.

We recruited the pregnant women between 12-20 gestational weeks at Obstetrics outpatient clinic in Ankara Gulhane Education and Research Hospital during routine antenatal care between May 2015 and March 2016. The eligibility criteria were as follows: having no major complication related to pregnancy and carrying at least one of the risk factors of preeclampsia discussed in the literature (American College of Obstetricians and Gynecologists, 2013; Bilano et al., 2014; Lisonkova and Joseph, 2013). The exclusion criteria included; having a miscarriage, unable to read or write in Turkish, moving to another city during the study, and changing the hospital for follow-ups or giving birth.

The sample size was calculated using the G Power 3.1.2 version computer package program according to the comparison of the self-efficacy-adequacy scale mean difference between the groups. So that 95% confidence interval and 80% power would be achieved as a mean size of effect, it was calculated that each group should consist of 45 pregnant women.

Randomization and Participation We selected totally 144 pregnant women at the beginning of the study. Later, 12 women did not meet eligibility criteria due to the diagnosis of pregnancy-related complications in the study period (five pregnant women dropped out of the study, and seven pregnant women planned to give birth in a different hospital). Finally, 132 pregnant women who met the eligibility criteria agreed to participate in this study and we randomized them as shown in Figure 1 Flow Chart. Eligible women were randomly allocated (ratio 1:1) into either a control group or study group following an allocation concealment process using an automatic computer-generated number table. After the randomization process, 13 pregnant women in control group and 19 pregnant women in study group were excluded from the study due to either moving to another city or having the miscarriage.

Ethics committee permission was obtained from the ethical committee of Ankara Gulhane Education and Research Hospital with the code 1491-2658-13/16484-303. As they involved human participants, all procedures were conducted in accordance with the ethical standards of the Declaration of Helsinki. We informed the women with risk of preeclampsia and who fulfilled the inclusion criteria about the study procedure, and obtained written informed consent.

Data collection The demographic information, obstetric and general health history were recorded for both groups at the first assessment. We applied Health Promoting Lifestyle Profile-II (HPLP II), the Self-Efficacy Scale (SES), pregnant and fetal follow-up forms 4 times during pregnancy. Finally, data of the women and their infants/newborn within postpartum 48 hours were collected.

In both groups, we recorded necessary information at every follow-up session within approximately 30 minutes (10 minutes for data collection for control & study group, 20 minutes for education and counseling for study group). We arranged first assessment and follow-up sessions between 12-20, 23-28, 29-34, 35-40 weeks of gestation.

The first version of the HPLP scale, was developed by Walker et al. in 1987 and revised in 1996 (Walker et al., 1987). The validity and reliability of the HPLP II in Turkish was tested by Bahar et al. and found to have a high level of validity and reliability (Bahar et al., 2008). The HPLP II questionnaire consist of 52 items and six dimensions, and it uses a four-point Likert scale from 1, indicating 'never', to 4, 'routinely'. Possible total scores on the questionnaire range from 52 to 208. Cronbach's alpha coefficient of the scale was 0.92.

The first version of the SES, developed by Shrer et al. in 1982 and the validity and reliability of the SES scale in Turkish was tested by Gozum and Aksayan in 1999 (Gözüm and Aksayan, 1999; Sherer et al., 1982). The SES consist of 23 items and uses a five-point Likert scale, in which 1 indicates "never defines me" and to 5, "defines me very well". Possible total scores on the questionnaire range from 23 to 115. Cronbach's alpha coefficient of the scale was 0.89.

We recorded the information, including presence of edema, feeling of movement of the baby, physical activity and breathing exercises in both groups on the pregnant and fetal follow-up form. In addition to these, we measured the blood pressure as well as non-stress test from the 34th gestation week. Pregnant women in the study group were asked to complete a daily follow-up form, recording their blood pressure, weight, edema, infant movement, and any problems. For each follow-up, the forms were collected and new forms were given and necessary reminders were made about regular filling.

Finally, after birth, in both groups maternal (preeclampsia development status, prenatal and postnatal blood pressure values and laboratory findings) and neonatal outcomes (first and fifth APGAR scores, baby's intensive care need, respiratory distress, birth weight and intra-uterine growth retardation) were collected with the postpartum data collection form, using information the women themselves, and information in their files.

Interventions Preeclampsia education and counseling program: We prepared a preeclampsia education booklet in accordance with the literature, (American College of Obstetricians and Gynecologists, 2013; Kasawara et al., 2012; Lisonkova and Joseph, 2013; You et al., 2012b). The content of the booklet was guided by the opinion of experts. It was written in easily understandable language and contained attractive and colorful illustrations. This booklet contents were definition and risk factors for the development of preeclampsia, maternal and fetal damages, recommendations for preventing its development (diet, rest, study, exercise, coping with stress techniques), follow-up of symptoms at home (blood pressure, weight and edema follow-up, counting fetal movements), danger signs, drug use, follow up in hospital, risk of developing in subsequent pregnancies, and its results. Pregnant women in the study group were given education and counseling at four times in addition to standard care, using the preeclampsia education booklet, in a special place. The participants' questions were answered, and each received a copy of the booklet. Pregnant women in the control group received standard prenatal care. Necessary reminders were made to attend regular follow-ups and their questions were answered during these. The researcher allowed participants to call her for consultations at any time.

Statistical analysis Data were analyzed using IBM SPSS version 22.0 (IBM Corp., Armonk, NY, USA) and p<0.05 was considered statistically significant. Descriptive statistics for the variables determined by counting; number and percentage (%); for the variables determined by measurement, mean±standard deviation (X ± SD), median and minimum-maximum (min-max) values were used. The conformity of continuous variables to normal distribution was evaluated by Kolmogorov Smirnov Test. To compare the groups for discrete variables; Chi-Square Test or Fisher Exact Test, for continuous variables; Student t Test or Mann-Whitney U Test were used. ANOVA was used for group comparisons for repeated measurements, and Bonferroni Test was used as post-hoc test. The error level was determined as 0.05 for all analyzes.

ELIGIBILITY:
* Having no major complication related to pregnancy
* Carrying at least one of the risk factors of preeclampsia discussed in the literature
* Being 12-20 gestational week
* Ability to read and write in Turkish,
* Volunteering to participate in the study.

Exclusion criteria:

* Having a miscarriage
* Unable to read or write in Turkish
* Moving to another city during the study
* Changing the hospital for follow-ups or giving birth.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-06-20 (Actual)

PRIMARY OUTCOMES:
maternal and neonatal health | an average of six months
  We used postpartum data collection form. After birth, in both groups maternal (preeclampsia development status, prenatal and postnatal blood pressure values and laboratory findings) and neonatal outcomes (first and fifth APGAR scores, baby's intensive care need, respiratory distress, birth weight and intra-uterine growth retardation) were collected with the postpartum data collection form, using information the women themselves, and information in their files.

SECONDARY OUTCOMES:
Health Promoting Lifestyle Profile-II (HPLP-II) | up to 22 weeks (4 times)
  We used Health Promoting Lifestyle Profile (HPLP) II scale. The first version of the HPLP scale, was developed by Walker et al. in 1987 and revised in 1996 (Walker et al., 1987). The validity and reliability of the HPLP II in Turkish was tested by Bahar et al. and found to have a high level of validity and reliability (Bahar et al., 2008).The HPLP II questionnaire consist of 52 items and six dimensions. These six subscales are nutrition, physical activity, spiritual growth, interpersonal relationship, health responsibility, and stress management. It uses a four-point Likert scale from 1, indicating 'never', to 4, 'routinely'. Possible total scores on the questionnaire range from 52 to 208. Cronbach's alpha coefficient of the scale was 0.92. Total score is directly proportional to healthy lifestyle behaviours.
Self-efficacy Scale (SES) | up to 22 weeks (4 times)
  We used self-efficacy scale (SES). The first version of the SES, developed by Shrer et al. in 1982 and the validity and reliability of the SES scale in Turkish was tested by Gozum and Aksayan in 1999 (Gözüm and Aksayan, 1999; Sherer et al., 1982).The SES consist of 23 items and uses a five-point Likert scale, in which 1 indicates "never defines me" and to 5, "defines me very well". Possible total scores on the questionnaire range from 23 to 115. Cronbach's alpha coefficient of the scale was 0.89.Total score is directly proportional to healthy lifestyle behaviours.

CONTACTS AND LOCATIONS:
Locations (1):
- Meltem Uğurlu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the study published in a journal

REFERENCES:
- [Background] Allen R, Rogozinska E, Sivarajasingam P, Khan KS, Thangaratinam S. Effect of diet- and lifestyle-based metabolic risk-modifying interventions on preeclampsia: a meta-analysis. Acta Obstet Gynecol Scand. 2014 Oct;93(10):973-85. doi: 10.1111/aogs.12467. PMID 25138651
- [Background] merican College of Obstetricians and Gynecologists, 2013. ACOG Guidelines: Hypertension in pregnancy, Washington, DC. https://doi.org/doi: 10.1097/01.AOG.0000437382.03963.88
- [Background] ACOG Committee Opinion No. 650: Physical Activity and Exercise During Pregnancy and the Postpartum Period. Obstet Gynecol. 2015 Dec;126(6):e135-e142. doi: 10.1097/AOG.0000000000001214. PMID 26595585
- [Background] Bilano VL, Ota E, Ganchimeg T, Mori R, Souza JP. Risk factors of pre-eclampsia/eclampsia and its adverse outcomes in low- and middle-income countries: a WHO secondary analysis. PLoS One. 2014 Mar 21;9(3):e91198. doi: 10.1371/journal.pone.0091198. eCollection 2014. PMID 24657964
- [Background] Blyton DM, Skilton MR, Edwards N, Hennessy A, Celermajer DS, Sullivan CE. Treatment of sleep disordered breathing reverses low fetal activity levels in preeclampsia. Sleep. 2013 Jan 1;36(1):15-21. doi: 10.5665/sleep.2292. PMID 23288967
- [Background] Gharaibeh M, Al-Ma'aitah R, Al Jada N. Lifestyle practices of Jordanian pregnant women. Int Nurs Rev. 2005 Jun;52(2):92-100. doi: 10.1111/j.1466-7657.2005.00257.x. PMID 15842321
- [Background] Kasawara KT, do Nascimento SL, Costa ML, Surita FG, e Silva JL. Exercise and physical activity in the prevention of pre-eclampsia: systematic review. Acta Obstet Gynecol Scand. 2012 Oct;91(10):1147-57. doi: 10.1111/j.1600-0412.2012.01483.x. Epub 2012 Jul 24. PMID 22708966
- [Background] Lange EM, Shah AM, Braithwaite BA, You WB, Wong CA, Grobman WA, Toledo P. Readability, content, and quality of online patient education materials on preeclampsia. Hypertens Pregnancy. 2015;34(3):383-90. doi: 10.3109/10641955.2015.1053607. Epub 2015 Jul 8. PMID 26153628
- [Background] Meles E, Giannattasio C, Failla M, Gentile G, Capra A, Mancia G. Nonpharmacologic treatment of hypertension by respiratory exercise in the home setting. Am J Hypertens. 2004 Apr;17(4):370-4. doi: 10.1016/j.amjhyper.2003.12.009. PMID 15062893
- [Background] Mol BWJ, Roberts CT, Thangaratinam S, Magee LA, de Groot CJM, Hofmeyr GJ. Pre-eclampsia. Lancet. 2016 Mar 5;387(10022):999-1011. doi: 10.1016/S0140-6736(15)00070-7. Epub 2015 Sep 2. PMID 26342729